CLINICAL TRIAL: NCT02384252
Title: Characterization of Obesity-related Cardiomyopathy Through Exploration of Human Atrial Trabeculae Contraction
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2012_09; 2012-A01605-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Heart Failure
Keywords: obese cardiomyopathy; mitochondria; contractile dysfunction
MeSH Terms: conditions — Obesity; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Right atrial tissue obtained during cannulation of the right atrium in preparation for cardiac surgery with extracorporeal circulation.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- obese patients: patients with BMI > 30
  Interventions: Other: functional tissu atrial analysis
- no obese patients: norma weight patient (BMI<25) overweight patients ( 25< BMI >30)
  Interventions: Other: functional tissu atrial analysis

INTERVENTIONS:
Other: functional tissu atrial analysis

SUMMARY:
The investigators aim to explore obese cardiomyopathy by studying contractile twitch force, sarcomere sensitivity to calcium and mitochondrial function in atrial myocardial samples of patients grouped according to their body mass index, i.e. normal weight, overweight and obese.

DETAILED DESCRIPTION:
Obesity is associated with the development of heart failure, regardless of coronary artery disease or other comorbidities.

Right atrial samples obtained from patients undergoing cardiac surgery and presenting no sign of clinical cardiomyopathy will be grouped according to patient's body mass index. Atrial trabeculae will be explored to dissect out the respective contribution of (i) sarcoplasmic reticulum dysfunction (isometric twitch force contraction analysis), (ii) abnormal sarcomere sensitivity to calcium assessed in permeabilized fibers and (iii) mitochondrial dysfunction to intrinsec contractile dysfunction of myocardium in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* patient schedulled for coronary artery bypass graft surgery or aortic valve replacement surgery with extracorporeal circulation
* must be over 18 years of age
* must be able to read and understand the consent form in French
* must be in sinus rhythm at inclusion time

Exclusion Criteria:

* medical history of type 1 diabetes
* medical history of sustained atrial arrhythmia
* pregnancy
* class III anti-arhythmic drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing coronary artery bypass graft surgery or aortic valve replacement surgery with extracorporeal circulation
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Intrinsic myocardial contractile force | the day of cardiac surgery
  twitch force developed by atrial trabeculae assessed in isometric conditions in atrial samples

SECONDARY OUTCOMES:
sarcomere sensitivity to calcium | the day of cardiac surgery
  force-calcium concentration relation assessed on permeabilized atrial fibers
Mitochondrial function | the day of cardiac surgery
  assesment of mitochondrial respiration and calcium retention capacity by oxygraphic measurement in saponin-permeabilized atrial fibers

CONTACTS AND LOCATIONS:
Overall Officials: David Montaigne, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Cardiologique - EFCV - CHRU, Lille, France